CLINICAL TRIAL: NCT04934332
Title: Early Ultrasound Screening of Heterotopic Ossification After Severe Neurological Trauma in a Post-intensive Care Rehabilitation Unit
Brief Title: Early Ultrasound Screening of Heterotopic Ossification After Severe Neurological Trauma
Acronym: POHER II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Paul Bennetot (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210785; IDRCB 2021-A01096-35 (Other: ANSM)
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Heterotopic Ossification
Keywords: heterotopic ossification; post intensive care rehabilitation unit; early screening; ultrasound; neurological trauma
MeSH Terms: conditions — Ossification, Heterotopic | interventions — High-Energy Shock Waves; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Newly hospitalized patients (Experimental): Patients admitted for the first time to a post intensive care rehabilitation unit after severe neurological trauma.
  Interventions: Procedure: Ultrasound; Procedure: CT scan; Procedure: Clinical examination

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound examination at 1 week and 5 weeks after admission.
Procedure: CT scan — CT scan at 5 weeks after admission. CT scan reader will be blinded to clinical data.
Procedure: Clinical examination — Weekly clinical examination from week-2 to week-5.

SUMMARY:
Prospective, bi-centric diagnostic, performance study on a new diagnostic procedure with ultrasounds against a reference diagnostic procedure.

The primary objective is to study the performance of ultrasound coupled with clinical examination at 1 week of admission for early screening of heterotopic ossification (HO) in patients admitted to a post intensive care rehabilitation unit (PICRU) after a severe neurologic trauma.

The CT scan at 5 weeks of admission is considered as the gold standard. CT scan reader will be blinded to clinical data.

DETAILED DESCRIPTION:
Heterotopic ossification still pose the problem of diagnosis and clinical management that is too late and invasive when complications arise. The challenge would be to identify patients at earlier stage of HO development in order to start an early treatment. This study will focus on the performance of ultrasound in the early screening of HO for patients admitted to a post intensive care rehabilitation unit after severe neurological trauma, this population being at high risk of HO.

Patient enrollment will be performed only at the PICRU of the Raymond Poincaré Hospital (AP-HP). Another center (the imaging department of the same hospital) will participate in this research for ultrasounds and CT scans, but will not perform any recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients ⩾ 18 years;
* Admitted to a neurological post intensive care rehabilitation unit for the first time;
* Hospitalized in ICU before being admitted to PICRU for a for traumatic brain injury (initial Glasgow coma scale < 14 and brain radiological abnormalities at the time of admission to ICU and / or a traumatic spinal cord injury (para- or tetraplegia with at least half of key muscles of the 2019 ISNCSCI classification with a strength of less than 3 below the neurological level of the injury at the time of admission to PICRU);
* Patient's written consent obtained (or from an authorized relative);
* Affiliation to a social security scheme.

Exclusion Criteria:

* History of moderate or severe traumatic brain injury;
* History of spinal cord injury (para- or tetraplegia);
* History of stroke or disabling neurological disease;
* History of hospitalization in neurological or neurosurgical or traumatological ICU for another reason;
* Breast-feeding or pregnancy;
* Under court protection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC (receiver operating characteristic) curve at 1 week | at 1 week
  Area under the ROC curve of ultrasound examination at 1 week compared CT scan at 5 weeks for making the diagnosis of HO.

SECONDARY OUTCOMES:
Sensitivity | at 1 week
  Sensitivity of ultrasound examination at 1 week for making the diagnosis of HO, the CT scan at 5 weeks of admission being considered as the gold standard.
Specificity | at 1 week
  Specificity of ultrasound examination at 1 week for making the diagnosis of HO, the CT scan at 5 weeks of admission being considered as the gold standard.
Positive predictive value and negative predictive value | at 1 week
  Positive predictive value and negative predictive value of ultrasound examination at 1 week for making the diagnosis of HO, the CT scan at 5 weeks of admission being considered as the gold standard.
Likelihood-ratio of ultrasound | at 1 week
  Likelihood-ratio of ultrasound examination at 1 week for making the diagnosis of HO, the CT scan at 5 weeks of admission being considered as the gold standard.
Area under the ROC curve at 5 weeks | at 5 weeks
  Area under the ROC curve of ultrasound examination at 5 weeks compared with CT scan at 5 weeks for making the diagnosis of HO.
Clinical examination | weekly from week-1 to week-5
  Area under the ROC curve of clinical examination at 1, 2, 3, 4, 5 weeks of admission compared with CT scan at 5 weeks to screen HO.

CONTACTS AND LOCATIONS:
Overall Officials: Julie PAQUEREAU, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France; Vincent T. CARPENTIER, MD, Study Director — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France
Locations (1):
- Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, Garche, France

IPD SHARING:
Plan to Share IPD: No